CLINICAL TRIAL: NCT03689426
Title: Using Cardiovascular Magnetic Resonance Tissue Characterisation and Wearable Technology to Predict Clinical Outcomes, Response to Therapy and Arrhythmias in Hospitalised Heart Failure Patients
Acronym: PREDICT-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CAR0540
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Heart Failure; Diffuse Fibrosis; Focal Fibrosis; Arrythmia
Keywords: Cardiovascular Magnetic Resonance Imaging; Tissue Characterisation; Wearable Technology; Prognosis; Response to Therapy
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma and urine samples will be stored for future 'OMICS' analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
150 patients admitted to University Hospital Southampton with heart failure will undergo comprehensive Cardiovascular Magnetic Resonance (CMR) imagining during their admission and continuous heart rhythm monitoring using wearable technology post discharge.

We hypothesise that analysis of this outcome data will discover novel CMR tissue characterisation and heart rhythm biomarkers that can be used to predict adverse clinical outcomes in heart failure populations and how individual patients will respond to specific therapies.

DETAILED DESCRIPTION:
PREDICT-HF a low risk single centre observational study in which 150 consecutive patients admitted with a new, primary diagnosis of heart failure undergo advanced CMR to non-invasively establish their individual myocardial tissue characteristics during their initial presentation.

All study participants will be invited to participate in an optional heart rhythm and rate monitoring sub study which will involve continuous electrocardiographic monitoring for up to 2 days prior to discharge and up to 30 day immediately post discharge using a Samsung S-PATCH device.

To enable multivariate statistical analysis to be performed each study participant will undergo a range of validated investigation to comprehensively establish and monitor other recognised heart failure prognostic biomarkers.

Participants will be managed per current NICE heart failure guidelines and will undergo rigorous clinical reviews at 6, 12 and 24 months. All clinically relevant event data e.g. MACE, rehospitalisation, decompensation and arrhythmias will be meticulously recorded for each participant throughout the study period.

This study will identify novel CMR derived tissue characterisation biomarkers of adverse outcome, response to therapy and arrhythmias in a hospitalised heart failure population. It will also be the first study to utilise wearable heart monitoring technology to accurately record heart rate and rhythm data in this population and investigate the potential impact of this on patient's clinical management and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* First hospital admission with a diagnosis of HF (as defined below)
* Able and willing to provide informed consent
* Able to undergo CMR

Exclusion Criteria:

* Known or subsequent diagnosis of amyloidosis, sarcoidosis or hypertrophic cardiomyopathy
* Severe valve disease of any type requiring inpatient surgery
* Heart transplant recipient or admitted for cardiac transplantation/ left ventricular assist device
* Clinically apparent myocardial ischemia which requires revascularisation
* Myocardial infarction or revascularisation within the previous 60 days
* Intra cardiac mass which requires surgery
* Active endocarditis
* Septicaemia
* Pregnancy
* Life expectancy <2 years secondary to any other cause (i.e. malignancy)
* Active treatment with chemotherapy
* Severe renal failure (GFR <30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted to University Hospital Southampton with a new primary diagnosis of heart failure will be considered for the study.
  The diagnosis of heart failure will be confirmed by a senior cardiologist with a subspecialty interest in heart failure following detailed review of the patient's history, clinical findings and investigations using the following diagnostic criteria:
  1. Signs and symptoms of heart failure
     &
  2. Objective evidence of cardiac dysfunction either by;
  Left ventricular ejection fraction of ≤ 50%
  or;
  Plasma concentrations of N-terminal pro-brain natriuretic peptide (NT-proBNP) >400 pg/mL if in sinus rhythm or > 1000 pg/ml if in atrial fibrillation/flutter and being treated with either oral or intravenous furosemide ≥40 mg/day or equivalent at the time of inclusion.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-04-30 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
All Cause Mortality | 2 years
  Number of deaths within the study population

SECONDARY OUTCOMES:
Rehospitalisation with heart failure | 2 years
  Number of Rehospitalisations with heart failure within the study population

OTHER OUTCOMES:
Cardiac arrythmia | 30 days
  The number of any cardiac arrhythmia following discharge within the study population

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided